CLINICAL TRIAL: NCT02955225
Title: Using Pressure Detecting Insoles to Reduce Knee Loading and Improve Function
Brief Title: Using Pressure Detecting Insoles to Reduce Knee Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF-6477
Record Dates: First submitted 2016-10-01; First posted 2016-11-04 (Estimated); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee loads; Knee adduction moment; Biomechanical intervention; Insole; Shoe
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexible shoe with Active Insole (Experimental): Subjects will be trained to change the plantar pressure using a flexible walking shoe with an activated pressure-detecting shoe insole (Moticon OpenGO insole).
  Interventions: Device: Active Moticon OpenGO insole
- Flexible shoe with Passive Insole (Active Comparator): A flexible walking shoe with a passive pressure-detecting shoe insole will be used for a comparator group.
  Interventions: Device: Passive shoe insole

INTERVENTIONS:
Device: Active Moticon OpenGO insole — A Moticon OpenGO insole measures shoe pressure and connects/sends data to a ANT+ enabled smartphone.
  Arms: Flexible shoe with Active Insole
Device: Passive shoe insole — A deactivated insole measures shoe pressure only.
  Arms: Flexible shoe with Passive Insole

SUMMARY:
The purpose of this study is to determine whether use of a pressure-detecting shoe improve can enhance favorable loading conditions at the knee.

DETAILED DESCRIPTION:
This is a randomized longitudinal proof-of-concept study. After a telephone prescreening, an in-person visit will screen for inclusion and exclusion criteria, requiring a clinical and radiographic assessment. A total of 40 subjects with symptomatic and radiographic medial knee OA will be enrolled in the study after obtaining informed consent. A total of three study visits will occur at the following time points: baseline, 3 weeks, and 6 weeks. At all three visits, the following outcome variables will be acquired: (1) joint loads during gait using 3D motion analysis and (2) knee symptoms, stiffness, pain, daily function, recreational function, and quality of life using the validated questionnaires. At the baseline visit, every participant will receive a standardized shoe and a pressure-detecting shoe insole. Randomly assigned to one of two groups, participants assigned to group A (n=25) will train for 3 weeks in the mobility shoe with active pressure-based feedback from the shoe insole, and group B (n=15) will train for three weeks in the mobility shoe with a passive shoe insole. All subjects will be encouraged to wear the study shoes containing the shoe insoles as their primary form of footwear and for a minimum of 6 hours/day, 6 days/week. They will be given a diary to record the daily time spent wearing the shoe/insole, daily analgesic history, and adverse events. These diaries will be reviewed at the 3 and 6 week study visits. After completing the third visit, subjects will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent and comply with the study protocol.
* Symptomatic OA of the knee greater than 3 months, as defined by the American College of Rheumatology's Clinical Criteria for Classification and Reporting of OA of the Knee. If symptoms are bilateral, then the knee identified as more symptomatic will serve as the index knee.
* Ambulatory knee pain, defined as the presence of greater than 30 mm of pain while walking on a flat surface (corresponding to question 1 of the visual analog format of the WOMAC).
* Radiographic OA of the study knee of grade 2 or 3, as defined by the modified Kellgren and Lawrence (K-L) grading scale.
* Medial compartment OA, defined as either qualitative joint space narrowing of ≥ 1or the presence of medial bone cyst, sclerosis, or osteophyte.
* Able to walk at least 10 minutes without a break.
* Age of 40 years or older

Exclusion Criteria:

* Unwillingness to wear study shoes for at least 6 hours/day for 6 days of the week
* Knee flexion contracture of > 15 degrees or inability to ambulate without assistance.
* Presence of clinical OA of the ankle or hip or ankle/hip pain>10 mm (WOMAC).
* Predominant lateral compartment OA, defined as narrowing of the lateral joint space in excess of the narrowing of the medial joint space in either knee.
* Concurrent systemic inflammatory arthropathy
* Prior knee or hip arthroplasty, or surgical arthroscopy within the previous 3 months.
* Intrinsic foot disease: hallux rigidus, hallux abducto-valgus, metatarsalgia, plantar fasciitis, peripheral neuropathy, or any foot condition that may be exacerbated particular footwear.
* Intra-articular knee injection: steroids within 6 wks, hyaluronan derivatives within 4 mos.
* Body mass index greater than 38.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10; Primary Completion 2021-08 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Wimmer, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be published through peer reviewed journals.
Supporting Information: Study Protocol
Time Frame: Dec 31, 2021
Access Criteria: Sharing access through the Arthritis Foundation

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole
Started | 26 | 12
Completed | 21 | 12
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole | Total
Number analyzed (Participants) | 26 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at the baseline visit
  years | 63 (9) | 63 (8) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 8 | 30
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 12 | 38
Knee Adduction Moment (KAM1) [Mean (Standard Deviation); unit: %bodyweight x height] — Surrogate marker of medial knee loading, measured using 3D motion analysis, with initial SI units in Newton*meters, and normalized to the individual's body weight and height, resulting in measurement units (% bodyweight * height).
  %bodyweight x height | 3.21 (0.99) | 3.27 (0.97) | 3.27 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Adduction Moment Relative to Baseline
Description: Surrogate marker of medial knee loading, measured using 3D motion analysis, with initial SI units in Newton*meters, and normalized to the individual's body weight and height, resulting in measurement units (% bodyweight * height).
  To assess changes in loading at the knee between baseline and the three post-baseline measurements (Immediately after initial training, after 3 weeks of ongoing training, after 6 weeks of ongoing training), participants underwent gait analysis in a motion analysis laboratory using force plates and optoelectric cameras to quantify the joint moments in three directions. This study focused on the change in joint moment in the frontal plane. After training with an active insole, we would expect reductions in the frontal plane knee joint moment. Generally speaking, lower moments are better and a negative change is desired.
Time Frame: Immediately after initial training, after 3 weeks of ongoing training, after 6 weeks of ongoing training
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of bodyweight x height
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole
Number analyzed (Participants) | 26 | 12
percentage of bodyweight x height
  Immediate | -0.21 [-0.31 to -0.11] | -0.09 [-0.24 to 0.07]
  3 weeks | -0.21 [-0.33 to -0.09] | -0.24 [-0.41 to -0.06]
  6 weeks (washout) | -0.12 [-0.24 to 0.01] | -0.12 [-0.35 to 0.01]

2. Secondary Outcome: Change in Moment Lever-arm for KAM
Description: To further assess changes in loading at the knee between baseline and the three post-baseline measurements (Immediately after initial training, after 3 weeks of ongoing training, after 6 weeks of ongoing training), participants underwent gait analysis in a motion analysis laboratory using force plates and optoelectric cameras to quantify joint moment. One component which determines the knee moment is the lever-arm between ground reaction force vector and the center of the knee joint, in the frontal plane, which is measured in millimeters.
Time Frame: Immediately after initial training, after 3 weeks of ongoing training, after 6 weeks of ongoing training
Measure: Least Squares Mean (95% Confidence Interval); unit: mm (millimeters)
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole
Number analyzed (Participants) | 26 | 12
mm (millimeters)
  Immediate | -6 [-9 to -4] | 1 [-3 to 4]
  3 weeks | -5 [-7 to -2] | 3 [-1 to 6]
  6 weeks (washout) | -2 [-4 to 1] | 3 [0 to 7]

3. Secondary Outcome: Change in SPEED
Description: A change in Speed (m/s) after 3 and 6 weeks of training with insoles.
Time Frame: Immediately after initial training, after 3 weeks of ongoing training, after 6 weeks of ongoing training
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters/sec
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole
Number analyzed (Participants) | 26 | 12
Meters/sec
  Immediate | -.09 [-.12 to -.05] | .05 [-.01 to .11]
  3 weeks | -.04 [-.09 to -.0] | .08 [.02 to .14]
  6 weeks (washout) | -.01 [-.06 to .03] | .06 [-.0 to .12]

4. Secondary Outcome: Change in Knee Pain
Description: To assess a change pain, participants completed the Knee Injury and Osteoarthritis Outcome Score (KOOS) at baseline, and after 3 and 6 weeks of training with insoles; 0 representing extreme problems and 100 representing no problems
Time Frame: after 3 weeks of ongoing training, after 6 weeks of ongoing training
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale from 0 to 100
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole
Number analyzed (Participants) | 26 | 12
units on a scale from 0 to 100
  3 week time point | 4.3 [-4.2 to 12.8] | 10.0 [-1.8 to 21.7]
  6 week time point | 7.0 [-4.2 to 18.2] | 12.3 [-2.7 to 27.3]

5. Secondary Outcome: Change in Self-reported Functional Status Between Baseline, After 3 Weeks of Training, and After 6 Weeks of Training
Description: To assess a change self-reported Functional status, participants completed the Knee Injury and Osteoarthritis Outcome Score (KOOS) at baseline, and after 3 and 6 weeks of training with insoles; 0 representing extreme problems and 100 representing no problems with Function in daily living, with a score of 100 as the optimal outcome with unlimited function. (change between baseline and 3 weeks, and the change between baseline and 6 weeks)
Time Frame: after 3 weeks of ongoing training, after 6 weeks of ongoing training
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale, from 0 to 100
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole
Number analyzed (Participants) | 26 | 12
units on a scale, from 0 to 100
  3 weeks | 8.5 [0.4 to 16.6] | 8.5 [-2.6 to 19.6]
  6 weeks | 15.6 [6.1 to 25.0] | 6.7 [-6.3 to 19.7]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Flexible Shoe With Active Insole | Flexible Shoe With Passive Insole
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/12
Other Adverse Events (participants affected / at risk) | 0/26 | 0/12

LIMITATIONS AND CAVEATS:
Since the goal of this proof-of-concept study was to evaluate feedback gait modification in individuals with knee OA, the study was primarily powered to determine KAM changes before and after the intervention and underpowered for comparison with another intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT02955225/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT02955225/SAP_001.pdf
  • Informed Consent Form (2020-07-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT02955225/ICF_002.pdf